CLINICAL TRIAL: NCT03308422
Title: Parental Representations of the Impact of the Use of Screens on Their Preschool Children Health and Development. An Opinion Survey of Parents of 1096 2-6-years-old Children
Brief Title: Parental Representations of the Impact of the Use of Screens on Their Preschool Children Health and Development.
Acronym: ECRENFANT
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: RNI2016/ECRENFANT-STEYER/YB
Record Dates: First submitted 2017-10-09; First posted 2017-10-12 (Actual); Last update posted 2017-10-12 (Actual); Status verified 2017-09

CONDITIONS: Parenting
Keywords: screens; preschool children; parenting education; social perceptions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parents of 2-6-years-old children: Parents of preschool children in Nancy agglomeration
  Interventions: Behavioral: parental representations

INTERVENTIONS:
Behavioral: parental representations — parental representations of the impact of the use of screens on their preschool children health and development

SUMMARY:
The main objective of this study was to evaluate the distribution of parental representations concerning the use of screens by preschool children, expressed in qualitative surveys: perceptions of screens as a source of learning, a source of appeasement, a source of behavioral difficulties and a source of reduction in the social interactions of young children.

The hypothesis of this study was the representations expressed in the qualitative studies were the reflection of the opinion of a majority of parents of young children.

ELIGIBILITY:
Inclusion Criteria:

* parents of 2-6-years-old preschool children

Exclusion Criteria:

* Minor parents

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parents of 2-6-years-old children educated in Nancy agglomeration
Sampling Method: Non-Probability Sample
Enrollment: 1096 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2017-04-07 (Actual); Study Completion 2017-04-07 (Actual)

PRIMARY OUTCOMES:
screens as a source of learning, of appeasement, of behavioral difficulties and of reduction in the social interactions of young children | baseline (J0)
  questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Dulong, Nancy, France